CLINICAL TRIAL: NCT00830648
Title: Safety of a Second Dose of Biken's Varicella Vaccine Administered at 4 to 6 Years of Age in Healthy Children in Argentina
Brief Title: Safety of a Second Dose of Biken's Varicella Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VBK12
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Varicella
Keywords: varicella-zoster virus; varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Live Attenuated Varicella Virus Vaccine

INTERVENTIONS:
Biological: Live Attenuated Varicella Virus Vaccine — 0.5 mL, Subcutaneous
  Other Names: Varicela Biken

SUMMARY:
The objective of the present study is to assess and document the safety of a second dose of Varicella Biken vaccine administered at 4 to 6 years of age in healthy children having previously received a first dose of Varicella Biken vaccine.

All subjects will receive a second dose of Varicella vaccine (Varicella Biken) at 4 to 6 years of age.

The expected total duration of follow-up (first visit to last visit) for each subject will be one month.

ELIGIBILITY:
Inclusion Criteria :

* Aged 4 to 6 years on the day of inclusion.
* Informed consent form signed by the parent(s) or legal guardian and by an independent witness.
* Subject and parent/guardian able to attend all scheduled visits and comply with all trial procedures.
* Written documentation of receipt of a first dose of Varicella Biken vaccine more than 3 months before inclusion.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances.
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the investigator.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination;
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination.
* Known Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen, or Hepatitis C seropositivity.
* History of varicella infection (confirmed either clinically, serologically or microbiologically).
* Previous vaccination against varicella disease with a vaccine different from Varicella Biken vaccine.
* Febrile illness (temperature ≥ 37.5°C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety after administration of Varicella vaccine | one month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Buenos Aires, Argentina

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com